CLINICAL TRIAL: NCT01521741
Title: Prospective Screening for Breast Cancer-related Lymphedema: Analysis of Objective Measurements, Symptoms, Functionality, and Quality of Life Questionnaires to Evaluate Lymphedema in Patients Following Treatment for Breast Cancer.
Brief Title: Prospective Screening for Breast Cancer-related Lymphedema
Status: Recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Alphonse Taghian, Chief of Breast Service, Massachusetts General Hospital
Other Study IDs: 08-540; R01CA139118 (NIH)
Record Dates: First submitted 2011-09-06; First posted 2012-01-31 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Lymphedema
Keywords: Breast Cancer; Lymphedema; Symptoms; Screening
MeSH Terms: conditions — Lymphedema; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Breast Cancer
  Interventions: Other: Breast Cancer-Related Lymphedema Screening

INTERVENTIONS:
Other: Breast Cancer-Related Lymphedema Screening — All patients enrolled in the trial will receive prospective BCRL screening from their pre-operative baseline throughout their breast cancer treatment process. All participants will be measured with perometry, bioimpedance spectroscopy, and patient-reported outcome measures.

SUMMARY:
The primary objectives of this study are twofold: 1) to detect and determine the level of symptoms, functional disability, and changes in quality of life that breast cancer patients experience from changes in their arms during and after treatment for breast cancer by collecting patient reported outcome measures, objective measurements, and clinical information in a prospectively maintained database and 2) to improve breast cancer-related lymphedema outcomes by early detection using objective measurements and symptoms assessments and assess these outcomes by maintaining the data in a database in order to contribute to the literature. The secondary aim of this study is to assess extracellular fluid content in the upper extremity, breast, and/or trunk of patients treated for breast cancer before, during, and after treatment in order to better understand the role of bioimpedance spectroscopy in lymphedema screening.

DETAILED DESCRIPTION:
The goal of the study is to create a large, prospectively maintained database with data from multiple objective measurement methods (i.e. perometry and BIS) that has detailed information on patient's symptoms and quality of life measures that can be used to answer research questions.

The study design is prospective in nature, and a questionnaire will be utilized in conjunction with objective measurements before, throughout, and after a patient's treatment for breast cancer. This protocol is designed to mimic the current standard of care screening program with the addition of the quality of life questionnaire and BIS measurements.

Data collection will include medical chart review, perometric arm volume measurements, BIS measurements, and a subjective questionnaire. At their preoperative multidisciplinary breast cancer clinic appointment, patients will undergo baseline arm volume measurements per standard of care. At this time, eligible patients will be offered this study. Those who consent will be given a baseline questionnaire to fill out and have baseline BIS measurements taken. Throughout their treatment and follow-up, patients will periodically have BCRL screening every 2-12 months depending on their risk (i.e. patients who are high risk for BCRL because of extensive lymph node surgery will be measured more often than patients who did not have lymph nodes removed). These screening visits will coincide with naturally occurring oncology follow-up visits; although, patients are also screened when patient or provider requests and questionnaires/BIS measurements will be offered at these time points as well.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of breast cancer
* Ability to obtain physical positioning for perometry (e.g. abducting shoulder to 90 degrees) and BIS measurements (e.g. standing without aid)

Exclusion Criteria:

* Evidence of distant metastatic disease that may cause edema,
* Previous breast cancer
* History of lymphedema
* Pregnancy at the time of accrual and/or cardiac implants (contraindications for BIS)
* Medical conditions that cause fluid retention or swelling (e.g. axillary cancer recurrence, renal insufficiency, congestive heart failure).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed breast cancer patients.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2009-08; Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Upper extremity changes following treatment for breast cancer | 1.5 to 5 years
  During and following treatment for breast cancer patients' experience a variety of changes in their upper extremities. The subject responses to the patient-reported outcome measures (BCLE-SEI questionnaire) obtained throughout their breast cancer treatment process will be analyzed in conjunction with arm volume measurements taken with both perometry and bioimpedance spectroscopy. This will allow for the correlation between quantifiable limb volume changes and subject documented changes in arm use and functionality and quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Alphonse G Taghian, MD PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ancukiewicz M, Miller CL, Skolny MN, O'Toole J, Warren LE, Jammallo LS, Specht MC, Taghian AG. Comparison of relative versus absolute arm size change as criteria for quantifying breast cancer-related lymphedema: the flaws in current studies and need for universal methodology. Breast Cancer Res Treat. 2012 Aug;135(1):145-52. doi: 10.1007/s10549-012-2111-8. Epub 2012 Jun 19. PMID 22710706
- [Background] Ancukiewicz M, Russell TA, Otoole J, Specht M, Singer M, Kelada A, Murphy CD, Pogachar J, Gioioso V, Patel M, Skolny M, Smith BL, Taghian AG. Standardized method for quantification of developing lymphedema in patients treated for breast cancer. Int J Radiat Oncol Biol Phys. 2011 Apr 1;79(5):1436-43. doi: 10.1016/j.ijrobp.2010.01.001. Epub 2010 Jun 3. PMID 20605339
- [Derived] Brunelle CL, Roberts SA, Horick NK, Gillespie TC, Jacobs JM, Daniell KM, Naoum GE, Taghian AG. Integrating Symptoms Into the Diagnostic Criteria for Breast Cancer-Related Lymphedema: Applying Results From a Prospective Surveillance Program. Phys Ther. 2020 Dec 7;100(12):2186-2197. doi: 10.1093/ptj/pzaa162. PMID 32931555